CLINICAL TRIAL: NCT05514847
Title: Low Dose Aspirin for Preterm Preeclampsia Prevention - a Randomized Trial of 81 Vs 162 Mg/day Dose in High-risk Patients
Brief Title: Low Dose Aspirin for Preterm Preeclampsia Preventionmg/day Dose in High-risk Patients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Christopher S. Ennen, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSR220148
Record Dates: First submitted 2022-08-16; First posted 2022-08-24 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-09

CONDITIONS: Preeclampsia; Pregnancy Related
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into 1 of 4 groups based on their results of two screening tests for preeclampsia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1 Control Group (No Intervention): Control Group (Group 1): These patients will be screened negative for both the ACOG screening test and the FMF preeclampsia screen. These women will receive no aspirin.
- 2 Randomized Group 1 (Active Comparator): Group 2: These patients will be screened negative for the ACOG screening test but positive for the FMF preeclampsia screen. These women will be randomized to either 81mg or 162 mg aspirin.
  Interventions: Drug: Aspirin 81Mg Ec Tab; Drug: Aspirin 162Mg Ec Tab
- 3 Standard of Care Group (Other): Group 3: These patients will be screened positive for the ACOG screening test but negative for the FMF preeclampsia screen. These women will be offered 81 mg aspirin, which is the standard of care.
  Interventions: Drug: Aspirin 81Mg Ec Tab
- Group 4 Randomized Group 2 (Active Comparator): Group 4: These patients will be screened negative for the ACOG screening test and positive for the FMF preeclampsia screen. These women will be randomized to either 81mg or 162 mg aspirin.
  Interventions: Drug: Aspirin 81Mg Ec Tab; Drug: Aspirin 162Mg Ec Tab

INTERVENTIONS:
Drug: Aspirin 81Mg Ec Tab — 81 mg enteric coated aspirin, taken daily from before 14 weeks of gestational age through pregnancy
  Arms: 2 Randomized Group 1; 3 Standard of Care Group; Group 4 Randomized Group 2
Drug: Aspirin 162Mg Ec Tab — 162 mg enteric coated aspirin, taken daily from before 14 weeks of gestational age through pregnancy
  Arms: 2 Randomized Group 1; Group 4 Randomized Group 2

SUMMARY:
This will be a randomized, open-label, controlled trial of patients at high risk of developing preeclampsia examining 81 mg/day vs 162mg/day daily acetylsalicylic acid (ASA) use. Based on screening results, patients will be randomized as outlined below into one of four groups. The proposed study is a pilot to determine if the higher dose of ASA has positive impacts on measures that predict preeclampsia, compared to the lower dose. If positive findings, data from this study could be used to develop a larger trial powered to determine if the higher ASA dose can improve clinical outcomes.

DETAILED DESCRIPTION:
This will be a randomized, open-label, controlled trial of patients at high risk of developing preeclampsia examining 81 mg/day vs 162mg/day daily ASA use. Currently, all patients that present to UVA Obstetric clinics are evaluated for development of preeclampsia per the current ACOG guidelines. If they screen positive per ACOG guidelines, then it is recommended they initiate 81mg/day ASA starting at 12 weeks of pregnancy and continuing until delivery. For this study, patients that present for early first trimester ultrasound (US) (for dating and/or genetic testing + ultrasound) will be offered enrollment in the study, and consenting patients will undergo double screening tests with ACOG and the FMF-based preeclampsia screen. This test will include first trimester uterine artery PI, assessment of maternal blood pressure, a maternal history and maternal serum markers including PAPP-A, PLGF, S-FLT, AFP. The first trimester preeclampsia screen will be performed between 10 weeks, 0 days and 13 weeks, 6 days of pregnancy.

For the patients within the intervention group, repeat uterine artery PI measurements will be performed during the patient's 20-week anatomic survey ultrasound. Repeat maternal serum biomarkers will be collected with routine 28-week labs and at time of delivery (standard times for blood draws in pregnancy) for all enrolled patients. Patients will be followed longitudinally through their pregnancy and delivery and neonatal outcomes will be recorded. Delivery and timing of delivery will be based solely on obstetric indications regardless of status in the trial. All uterine artery Doppler measurements will be obtained by P.J. Kumar.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Ages 18-50
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Pregnant female in the first trimester.
* Ability to take oral medication and be willing to adhere to the aspirin regimen
* Patient has a prenatal ultrasound between 11+0 through 13+6 days of gestation
* Patient who has low or high risks for preeclampsia by the ACOG (American College of Obstetricians and Gynecologists) screening tool, and low or high risks for the FMF prescreening tool for preeclampsia.

Exclusion Criteria:

* ASA allergy, known hypersensitivity to NSAIDS
* Patients with nasal polyps
* Patients with aspirin-induced asthma exacerbations
* Active peptic ulcer disease
* Severe hepatic dysfunction
* History of GI bleeding
* Pregnancy with major abnormalities demonstrated on the 11-13-week scan
* Patient presents beyond 13w6d for first prenatal visit
* Age < 18
* Non-viable pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must be pregnant
Enrollment: 150 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The impact of 81mg/day vs 162 mg/day aspirin on PAPP-A | from before 14 weeks gestation age through delivery (up to 41 weeks gestation)
  To assess the effect of 81mg/day vs 162mg/day on the progression of PAPP-A in pregnancy. Unit of measure is multiples of the median (MoM).
The impact of 81mg/day vs 162 mg/day aspirin on PGLF (Placenta growth factor) | from before 14 weeks gestation age through delivery (up to 41 weeks gestation)
  To assess the effect of 81mg/day vs 162mg/day on the progression of PGLF in pregnancy. Unit of measure is multiples of the median (MoM).
The impact of 81mg/day vs 162 mg/day aspirin on S-FLT | from before 14 weeks gestation age through delivery (up to 41 weeks gestation)
  To assess the effect of 81mg/day vs 162mg/day on the progression of S-FLT in pregnancy. Unit of measure is multiples of the median (MoM).
The impact of 81mg/day vs 162 mg/day aspirin on AFP (alpha fetal protein) | from before 14 weeks gestation age through delivery (up to 41 weeks gestation)
  To assess the effect of 81mg/day vs 162mg/day on the progression of AFP in pregnancy. Unit of measure is multiples of the median (MoM).

SECONDARY OUTCOMES:
The impact of 81 mg/day vs 162 mg/day aspirin dosage on Uterine artery pulsatility average in patients with 81 vs 162 mg/day of ASA | from before 14 weeks gestation age through delivery (up to 41 weeks gestation)
  The uterine artery pulsaltility index will be reviewed. This will be obtained via doppler ultrasound studies This will be described on a continuous scale with repeated measures and analyzed using T-test and ANOVA. Uterine artery doppler pulsatile index (PI) will be measured in the first, second and third trimester of pregnancy using doppler mode on the ultrasound
  We will use these data to determine the ability to predict adverse outcomes by uterine artery Doppler parameters and mean arterial pressure. We predict that the uterine artery PI will be lower in the 162mg/day group compared to the 81mg/day group. Furthermore, uterine artery PI will increase in those that are at high risk of developing PE compared to the control group.
The impact of 81 mg/day vs 162 mg/day aspirin on maternal outcomes | from before 14 weeks gestation age through delivery and resolution of any pregnancy and delivery-related illnesses (up to 6 weeks postpartum)
  Maternal outcomes including:
  * Mode of delivery
  * Antepartum stillbirth
  * Pre-pregnancy medical conditions
  * hemorrhage
  * Abruption
  * Development of fetal growth restriction (FGR)
  * Develop of hypertensive disorder of pregnancy
  * Post-partum blood pressure and medication adjustments
  * oligohydramnios, polyhydramnios,
  * gestational age at delivery
  * blood pressure at delivery
  * labor course including need for magnesium
The impact of 81 mg/day vs 162 mg/day aspirin on fetal outcomes | from before 14 weeks gestation age through discharge from hospital following delivery (up to 6 weeks post birth)
  Fetal outcomes including:
  * Gestational age (GA) at time of delivery
  * Neonatal intensive care unit (NICU) length of stay
  * Estimated fetal weight compared to birth weight
  * Intrapartum stillbirth
  * Need for fetal interventions including: mechanical ventilation, CPAP
  * Apgar scores at 1,5 minutes
  * Arterial cord pH
  * Intraventricular hemorrhage (IVH), Necrotizing enterocolitis (NEC), sepsis, neonatal death, neonatal seizures, neonatal end organ dysfunction, fetal anemia

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Kumar, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No